CLINICAL TRIAL: NCT04353609
Title: Covid-19 in Patients With Chronic Inflammatory Rheumatism, Auto-immune or Auto-inflammatory Rare and Non-rare Diseases : a Retrospective Multicenter Observational Study
Brief Title: Covid-19 in Patients With Chronic Inflammatory Rheumatism, Auto-immune or Auto-inflammatory Rare and Non-rare Diseases
Acronym: covid19 fai2r
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: FAI²R (Auto-immune and auto-inflammatory rare diseases French network) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI_2020_03
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2; Chronic Inflammatory Rheumatism; Autoimmune Diseases
Keywords: Covid-19; chronic inflammatory rheumatism; auto-immune diseases; auto-inflammatory diseases; intensive care unit
MeSH Terms: conditions — Autoimmune Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since December 2019, an international outbreak of respiratory illnesses caused by SARS-CoV-2 called covid-19 has become a global challenge. In France, while the first cases were reported in January, more than 20 000 cases were confirmed at end of March. Early estimations from epidemiological data seem to show that 18-20% of patients with confirmed covid-19 are admitted in an intensive care unit (ICU). Patients with chronic inflammatory rheumatism, auto-immune or auto-inflammatory rare and non-rare diseases are susceptible to severe covid-19 (i.e ICU) due to the specific therapeutic management of their illness (corticosteroid, immunosuppressive and immunomodulatory drugs,..). No data are available for this particular population in France.

This retrospective multicentre observational study aims to evaluate the frequency of severe forms of covid-19 and risk factors associated with specific outcomes in covid-19 in patients with chronic inflammatory rheumatism, auto-immune or auto-inflammatory rare and non-rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients, children and adults
* Patients with known chronic inflammatory rheumatism, auto-immune or auto-inflammatory rare and non-rare diseases with proven/suspected SARS-Cov-2 infection (COVID-19) (by biological data (serological or positive Cov-2 PCR) or CT scan images or clinical observations consistent with covid-19)

Exclusion Criteria:

* patients opposed to the use of their data
* patients under guardianship, protected persons

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with chronic inflammatory rheumatism, auto-immune or auto-inflammatory rare and non-rare diseases with proven SARS-Cov-2 infection (COVID-19) taken care in hospital or in private practice by rheumatologist, internist or pediatrician working in both hospital and private practice activities
Sampling Method: Non-Probability Sample
Enrollment: 13770 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients presenting a severe form of covid-19 requiring an intensive care unit admission or leading to death | From Baseline up to Day 21 after first symptoms of covid-19

SECONDARY OUTCOMES:
Proportion of patients who die from a severe form of covid-19 | From Baseline up to Day 21 after first symptoms of covid-19
Proportion of patients who present an history of diabetes according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present obesity (validated by Body Mass Index value > 30 kg/cm2) | At the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of Chronic Pulmonary Obstructive Disease according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of Asthma according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of Hypertension according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of cardiac disease according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of Pulmonary Interstitial Disease according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of stroke according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of angiotensin-converting-enzyme inhibitor according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)
Proportion of patients who present an history of cancer according to medical records | Before the set-up of first symptoms of covid-19 (Baseline visit)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hachulla, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrot L, Boyer L, Flipo RM, Marotte H, Pertuiset E, Miceli C, Thomas T, Seror R, Chazerain P, Roux N, Richez C, Pham T; FAI2R/SFR/SNFMI/SOFREMIP/CRI/IMIDIATE consortium. Factors associated with COVID-19 severity in patients with spondyloarthritis: Results of the French RMD COVID-19 cohort. Joint Bone Spine. 2023 Dec;90(6):105608. doi: 10.1016/j.jbspin.2023.105608. Epub 2023 Jul 5. PMID 37414137
- [Derived] Truchetet ME, Drumez E, Barnetche T, Martin C, Devaux M, Goulenok T, Maria A, Schmidt J, Abdallah NA, Melki I, Hachulla E, Richez C. Outcome of COVID-19 in patients with rheumatic and inflammatory diseases treated with mycophenolic acid: data from the French RMD COVID-19 cohort. RMD Open. 2022 Sep;8(2):e002476. doi: 10.1136/rmdopen-2022-002476. PMID 36113962
- [Derived] Avouac J, Drumez E, Hachulla E, Seror R, Georgin-Lavialle S, El Mahou S, Pertuiset E, Pham T, Marotte H, Servettaz A, Domont F, Chazerain P, Devaux M, Claudepierre P, Langlois V, Mekinian A, Maria ATJ, Banneville B, Fautrel B, Pouchot J, Thomas T, Flipo RM, Richez C; FAI2R/SFR/SNFMI/SOFREMIP/CRI/IMIDIATE consortium and contributors; FAIR/SFR/SNFMI/SOFREMIP/CRI/IMIDIATE consortium and contributors. COVID-19 outcomes in patients with inflammatory rheumatic and musculoskeletal diseases treated with rituximab: a cohort study. Lancet Rheumatol. 2021 Jun;3(6):e419-e426. doi: 10.1016/S2665-9913(21)00059-X. Epub 2021 Mar 25. PMID 33786454
- [Derived] FAI2R /SFR/SNFMI/SOFREMIP/CRI/IMIDIATE consortium and contributors. Severity of COVID-19 and survival in patients with rheumatic and inflammatory diseases: data from the French RMD COVID-19 cohort of 694 patients. Ann Rheum Dis. 2021 Apr;80(4):527-538. doi: 10.1136/annrheumdis-2020-218310. Epub 2020 Dec 2. PMID 33268442